CLINICAL TRIAL: NCT04019132
Title: Power During Functional Tasks in Older Adults: Reliability, Reference Values and Relationship With Other Outcome Measurements Related to Sarcopenia
Brief Title: Power During Functional Tasks in Older Adults
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S62540
Record Dates: First submitted 2019-07-02; First posted 2019-07-15 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Aging
Keywords: Muscle Power; Functional capacity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Older adults: Older adults aged >65 years
  Interventions: Diagnostic Test: Muscle function test
- Young group: Younger adults between the age of 20 and 40 years
  Interventions: Diagnostic Test: Muscle function test
- Middle-aged group 1: Adults between the age of 40 and 55 years
  Interventions: Diagnostic Test: Muscle function test
- Middle-aged group 2: Adults between the age of 55 and 65 years
  Interventions: Diagnostic Test: Muscle function test

INTERVENTIONS:
Diagnostic Test: Muscle function test — Body measurements, power and strength tests of the knee extensor muscle, handgrip strength, functional capacity tests, objective measurement of physical activity (subgroup of older adults, n=50)

SUMMARY:
The primary aim of this study is to optimize the methodology to measure lower limb power in older adults, so that clinicians are able to detect functional problems in this population earlier.

DETAILED DESCRIPTION:
Aging is associated with slower movement patterns, a higher fall risk and a restriction in functionality. This will lead to an increase in the number of dependent elderly and a high socio-economic burden. From the age of 40, a systematic loss of muscle mass and muscle force, also known as sarcopenia, will occur. In addition, performing daily tasks requires the production of muscle force at a certain speed. The product of force and speed, power, decreases even earlier and faster than muscle force.

This power is typically measured with specialized equipment, which limits the large-scale applicability. With the help of accelerometry there is the possibility to measure power during more functional tasks and movements, which benefits the applicability, but the reliability, reference values and link with other outcome measurements related to sarcopenia has to be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Age >20

Exclusion Criteria:

* Unstable cardiovascular diseases
* Fever or acute infection
* Cognitive or physical malfunctioning that hinders the understanding or performance of tests and/or instructions

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy young to older adults
Sampling Method: Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Lower limb muscle power during a stair climb test | 1 test moment of approximately 1 hour, planned between September 2019 and July 2020
  The power (watt) needed to perform stair climbing is calculated using a 3D accelerometer (DynaPort MoveTest, McRoberts), worn at the back of the participant
Lower limb muscle power during a sit-to-stand test | 1 test moment of approximately 1 hour, planned between September 2019 and July 2020
  The power (watt) needed to perform 5 sit-to-stand transitions and a 30 sec. sit-to-stand test is calculated using a 3D accelerometer (DynaPort MoveTest, McRoberts), worn at the back of the participant
Reliability of power measurements measured with a 3D accelerometer | 1 test moment of approximately 30 minutes, planned between September 2019 and July 2020
  Reliability of power measurements (watt) measured with a 3D accelerometer (DynaPort MoveTest, McRoberts) worn during functional activities (stair climbing, sit-to-stand test) three times within a period of 2 weeks
Rate of power (force-velocity) development | 1 test moment of approximately 1 hour, planned between September 2019 and July 2020
  Participants perform a test protocol on a Biodex Dynamometer. The rate of power development (watt/s) is defined as the linear slope of the power-time curve and is measured from the onset of movement till peak power.
Handgrip strength | 1 test moment of approximately 1 hour, planned between September 2019 and July 2020
  Handgrip strength (kg) evaluated with a Jamar dynamometer
Jumping height | 1 test moment of approximately 1 hour, planned between September 2019 and July 2020
  Jumping height (in cm) measured during a standardized jump test
Physical activity | 1 week
  Objective measurement of physical activity in a subgroup of older participants (n=50) by means of accelerometry
Number of steps/stairs a day | 1 week
  Objective measurement of physical activity in a subgroup of older participants (n=50) by means of accelerometry

SECONDARY OUTCOMES:
Number of repetitions during a 30s sit-to-stand test | 1 test moment of approximately 1 hour, planned between September 2019 and July 2020
  Number of complete sit-to-stand transitions in 30 sec.
6min walk distance | 1 test moment of approximately 1 hour, planned between September 2019 and July 2020
  The walk distance (in m) covered in 6 min.
Balance | 1 test moment of approximately 1 hour, planned between September 2019 and July 2020
  Number of seconds a participant can hold a tandem stand, a semi-tandem stand or with the feet together
Maximal gait speed | 1 test moment of approximately 1 hour, planned between September 2019 and July 2020
  The average speed to walk 3m as fast as possible (in m/s)
Usual gait speed | 1 test moment of approximately 1 hour, planned between September 2019 and July 2020
  The average speed to walk 4m at a usual pace (in m/s)
Maximal isometric strength | 1 test moment of approximately 1 hour, planned between September 2019 and July 2020
  Maximal strength (Nm) is measured by means of unilateral isometric knee-extensor tests on a Biodex Dynamometer
Maximal isokinetic strength | 1 test moment of approximately 1 hour, planned between September 2019 and July 2020
  Maximal strength (Nm) is measured by means of unilateral isokinetic knee-extensor tests on a Biodex Dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven - Department of Movement Sciences, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No